CLINICAL TRIAL: NCT00304187
Title: Effects of Erythromycin on Binge Eating and GI Function in Bulimia Nervosa
Brief Title: Effectiveness of Antibiotic Treatment for Reducing Binge Eating and Improving Digestive Function in Bulimia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, B. Timothy Walsh, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #4902; R01MH042206-05 (NIH); DATR A2-AID (Other: NIH Adult Translational Research and Treatment Development)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-06

CONDITIONS: Bulimia Nervosa; Eating Disorders
Keywords: Binge-Eating Disorder
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders; Binge-Eating Disorder | interventions — Erythromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythromycin (Experimental): Subjects with Bulimia Nervosa will take erythromycin.
  Interventions: Drug: Erythromycin
- Placebo (Placebo Comparator): Participants will take matched placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythromycin — Erythromycin, 250 mg or 500 mg, three times a day for 6 weeks
  Other Names: E-mycin; Eryc; Ery-tab
  Arms: Erythromycin
Drug: Placebo — Placebo, 250 mg or 500 mg, three times a day for 6 weeks
  Other Names: inactive substance
  Arms: Placebo

SUMMARY:
This study will determine the effectiveness of the antibiotic erythromycin in enhancing gastrointestinal function and decreasing the frequency of binge eating in people with bulimia nervosa.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is a serious eating disorder that is characterized by frequent uncontrolled eating binges. These binges are often followed by compensatory behavior, including the following: self-induced vomiting; misuse of laxatives, diuretics, enemas, or other medications to induce purging; fasting; or excessive exercise. If left untreated, BN can lead to many serious health issues: tooth decay; irregular menstruation; bowel damage; constipation; heart and kidney disease; intestinal damage; puffiness, especially in the face and fingers; increased hair growth on the face and body; and mineral imbalances in the body. Although there is significant existing knowledge about the characteristics and treatment of BN, more information is needed about gastrointestinal (GI) function and its effect on binge eating behavior. This study will determine the effectiveness of the antibiotic erythromycin in enhancing GI function and decreasing the frequency of binge eating in people with BN.

Participants in this 8-week, double-blind study will first undergo gastric emptying and GI hormone release testing for 1 day. Within 1 week of completing these pre-treatment tests, participants will be randomly assigned to receive either erythromycin or placebo for 6 weeks. Upon medication assignment, participants will meet with a psychiatrist to receive their assigned medication. Participants will receive medication at weekly study visits. Medication dosage will be increased if symptoms do not improve, or decreased if adverse medication side effects are reported. A final day of gastric emptying and GI hormone release testing, as well as routine blood tests, will take place in Week 7, after 6 weeks of medication treatment. Participants' weight will be measured at Weeks 1, 4, and 7. Participants will also receive an EKG 1 week after each upward dosage adjustment. Patients will be informed of their medication assignment at the Week 7 study visit, and will be referred to a non-study clinician for further treatment.

For information on related studies, please see NCT00308776 and NCT00307190.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for bulimia nervosa
* Duration of illness is greater than 1 year
* Self-induces vomiting
* Weighs 80%-120 % of ideal weight

Exclusion Criteria:

* Significant medical illness
* Current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder, as defined by American Psychiatric Association criteria
* Moderate to severe depression, as defined by a score greater than 18 on the Hamilton Depression Scales
* Current diagnosis of organic mental disorder, factitious disorder, or malingering
* History of a personality disorder (e.g., schizotypal, borderline, or antisocial) that might interfere with assessment or compliance with the study procedures
* At risk for suicide
* Current psychotropic medications and current medications that affect GI function or that inhibit or induce cytochrome three A gene expression
* Currently pregnant, lactating, or planning to become pregnant
* Drug or alcohol abuse within the 3 months prior to study entry
* Abnormal EKG at baseline or 1 week following each upward dosage adjustment
* Anemia
* Known intolerance to erythromycin, or related antibiotics
* Abnormal results on liver function tests
* Electrolyte abnormalities

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2004-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. T. Walsh, MD, Principal Investigator — New York State Psychiatric Institute at Columbia University Medical Center
Locations (1):
- Eating Disorders Clinic, New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eating Disorders Research Clinic at New York State Psychiatric Institute
Groups:
- Erythromycin: Subjects with Bulimia Nervosa will take erythromycin.
  Erythromycin : Erythromycin, 250 mg or 500 mg, three times a day for 6 weeks
- Placebo: Participants will take matched placebo.
  Placebo : Placebo, 250 mg or 500 mg, three times a day for 6 weeks
Period: Overall Study
Arm/Group | Erythromycin | Placebo
Started | 15 | 14
Completed | 13 | 13
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythromycin | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (3) | 24 (3) | 24 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Binge Frequency
Description: Binge frequency was assessed by patient diary. All patients were asked to keep a diary of the number of daily binge eating and vomiting episodes which was collected at each weekly visit.
Time Frame: Measured at Week 7
Population: Participants for analysis included 13 patients in the erythromycin and 13 patients in the placebo group who completed at least 5 weeks of drug treatment.
Measure: Mean (Standard Deviation); unit: Binge Episodes/Week
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 13 | 13
Binge Episodes/Week | 10.4 (8.7) | 11.3 (10.9)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority; p < .05, t-test, 2 sided

2. Primary Outcome: Percent of Meal Remaining/Minute
Description: percent of meal remaining/minute
Time Frame: Measured at Week 7
Measure: Mean (Standard Error); unit: percent of meal remaining/minute
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 13 | 13
percent of meal remaining/minute | -.339 (.14) | -.177 (.122)

ADVERSE EVENTS:
Arm/Group | Erythromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No